CLINICAL TRIAL: NCT01181869
Title: Observatoire de l'ANTADIR - Database of Patients Registered as Treated With Respiratory Support in a Multicenter Homecare Federation for Patients Wirh Respiratory Problems
Brief Title: Database of Patients Treated With Respiratory Support
Acronym: observatory
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Principal Investigator, Daniel VEALE, Investigator, Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Other Study IDs: observatoire antadir; 1983 (Other: antadir)
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Respiratory Failure
Keywords: respiratory failure; oxygen; sleep apnoea; ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Sleep Apnea Syndromes; Respiratory Aspiration | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Oxygen therapy: Database of patients on oxygen
  Interventions: Device: oxygen
- ventilation: database of patients on ventilatory support
  Interventions: Device: oxygen
- Continuous positive airway pressure: Sleep apnoea patients on CPAP
  Interventions: Device: oxygen

INTERVENTIONS:
Device: oxygen — oxygen therapy, ventilation for respiratory failure CPAP for sleep apnoea
  Other Names: LTOT; NIV; CPAP

SUMMARY:
An observatory of patients registered in 22 local homecare associations in France, for respiratory diseases, with annual data update. Demographic and clinical data are registered rendering possible extraction of clinical and prognostic data.

DETAILED DESCRIPTION:
Patients on treatment for respiratory failure and for sleep apnoea are registered on entry into treatment with recording of clincal and demographic data. Data available on age, sex, region, respiratoy function, blood gases, smoking status and some bilogical data

ELIGIBILITY:
Inclusion Criteria:

* requiring respiratory support

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring respiratory support, in the ANTADIR homecare federation
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 1983-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
death | 20 years
  long term follow up of a regularly updated database

SECONDARY OUTCOMES:
treatment adjustment | 20 years
  Change of treatment from oxygen to ventilatioion or other evolution

CONTACTS AND LOCATIONS:
Overall Officials: Daniel VEALE, MD, Study Director — ANTADIR scientific committee; Jean Francois MUIR, MD, Study Chair — Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Locations (1):
- ANTADIR, Paris, France

REFERENCES:
- [Result] Chambellan A, Chailleux E, Similowski T; ANTADIR Observatory Group. Prognostic value of the hematocrit in patients with severe COPD receiving long-term oxygen therapy. Chest. 2005 Sep;128(3):1201-8. doi: 10.1378/chest.128.3.1201. PMID 16162707
- [Result] Chailleux E, Laaban JP, Veale D. Prognostic value of nutritional depletion in patients with COPD treated by long-term oxygen therapy: data from the ANTADIR observatory. Chest. 2003 May;123(5):1460-6. doi: 10.1378/chest.123.5.1460. PMID 12740261
- [Result] Chailleux E, Boffa C. [Chronic respiratory insufficiency in France]. Rev Prat. 2001 May 31;51(10):1061-5. French. PMID 11468903
- [Result] Veale D, Chailleux E, Hoorelbeke-Ramon A, Reybet-Degas O, Humeau-Chapuis MP, Alluin-Aigouy F, Fleury B, Jonquet O, Michard P. Mortality of sleep apnoea patients treated by nasal continuous positive airway pressure registered in the ANTADIR observatory. Association Nationale pour le Traitement A Domicile de l'Insuffisance Respiratoire chronique. Eur Respir J. 2000 Feb;15(2):326-31. doi: 10.1034/j.1399-3003.2000.15b18.x. PMID 10706500
- [Result] Veale D, Chailleux E, Taytard A, Cardinaud JP. Characteristics and survival of patients prescribed long-term oxygen therapy outside prescription guidelines. Eur Respir J. 1998 Oct;12(4):780-4. doi: 10.1183/09031936.98.12040780. PMID 9817145
- [Result] Voisin C. [Medico-social management of severe respiratory insufficiency. Role of Associations]. Bull Acad Natl Med. 1998;182(6):1159-71; discussion 1172. French. PMID 9812404
- [Result] Chailleux E, Fauroux B, Binet F, Dautzenberg B, Polu JM. Predictors of survival in patients receiving domiciliary oxygen therapy or mechanical ventilation. A 10-year analysis of ANTADIR Observatory. Chest. 1996 Mar;109(3):741-9. doi: 10.1378/chest.109.3.741. PMID 8617085
- See also: ANTADIR website — http://antadir.com